CLINICAL TRIAL: NCT05266690
Title: Effect of Degree of Polymerization and Linkage of α-glucans on Post-prandial Glucose Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 19.10.NRC
Record Dates: First submitted 2022-02-07; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Postprandial Glucose Response
Keywords: Postprandial glucose response; α-glucans; Polymerization; Decentralized study design

STUDY DESIGN:
Intervention Model Description: Monocentric, controlled, randomized, double-blind, complete 4x4 cross-over clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Individual coding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sequence 1 (Experimental): Roquette Glucidex 40 - Roquette Glucidex 2 - Pharmacosmos Dextran 10 - Promitor 70
  Interventions: Dietary Supplement: Roquette Glucidex 2; Dietary Supplement: Pharmacosmos Dextran 10; Dietary Supplement: Roquette Glucidex 40; Dietary Supplement: Promitor 70
- Sequence 2 (Experimental): Roquette Glucidex 2 - Promitor 70 - Roquette Glucidex 40 - Pharmacosmos Dextran 10
  Interventions: Dietary Supplement: Roquette Glucidex 2; Dietary Supplement: Pharmacosmos Dextran 10; Dietary Supplement: Roquette Glucidex 40; Dietary Supplement: Promitor 70
- Sequence 3 (Experimental): Promitor 70 - Pharmacosmos Dextran 10 - Roquette Glucidex 2 - Roquette Glucidex 40
  Interventions: Dietary Supplement: Roquette Glucidex 2; Dietary Supplement: Pharmacosmos Dextran 10; Dietary Supplement: Roquette Glucidex 40; Dietary Supplement: Promitor 70
- Sequence 4 (Experimental): Pharmacosmos Dextran 10 - Roquette Glucidex 40 - Promitor 70 - Roquette Glucidex 2
  Interventions: Dietary Supplement: Roquette Glucidex 2; Dietary Supplement: Pharmacosmos Dextran 10; Dietary Supplement: Roquette Glucidex 40; Dietary Supplement: Promitor 70

INTERVENTIONS:
Dietary Supplement: Roquette Glucidex 2 — Roquette Glucidex 2: Maltodextrins with high degree of polymerization
Dietary Supplement: Pharmacosmos Dextran 10 — Pharmacosmos Dextran 10: Dextran with high degree of polymerization
Dietary Supplement: Roquette Glucidex 40 — Roquette Glucidex 40: Glucose syrup
  Other Names: Positive control
Dietary Supplement: Promitor 70 — Promitor 70: Resistant Dextrin with a complex structure containing 70% non-digestible dietary fiber
  Other Names: Negative control

SUMMARY:
The primary research project objective is to investigate whether a maltodextrin with high degree of polymerization (Roquette Glucidex 2) and a dextran with comparable degree of polymerization (Pharmacosmos Dextran 10) have lower post-prandial glucose response than glucose syrup (Roquette Glucidex 40). To confer further robustness to the results, the post-prandial glucose response will be compared to a negative control represented by a resistant dextrin with a complex structure containing 70% non-digestible dietary fiber (Promitor 70), which is currently used for sugar replacement.

Additional key objective is to investigate the safety and gastrointestinal tolerability of the investigational products.

DETAILED DESCRIPTION:
The aim of the present research project is to generate comparative data on post-prandial glucose response (PPGR) of α-glucans varying systematically degree of polymerization and linkage type. These data are expected to contribute to the sugar replacement strategy in food industry.

An additional goal of the study is to demonstrate the feasibility of running a PPGR study remotely, i.e. with the participants carrying out most of the procedures at home.

Remote clinical trials (so called "virtual") have recently started to be implemented in pharmaceutical clinical research with the intent to reduce the burden on participants and investigational sites, narrow gaps with real life conditions, expand recruitment potential and maximize data collection. Nutritional research could be an even more suitable context for the remote approach because of the much lower safety risks for the participants.

However, with this innovative approach come new risks (at distance communication with the participants, complex data flows and logistics, lower degree of control on clinical trial execution) that can potentially affect the reliability of the study results and therefore require proper mitigation.

In the present study the following measures were put in place to reduce those risks:

* Clear and complete instructions will be provided to the subjects on how the carry out remotely the study procedures.
* Digital tools and devices used for data capture will be easy to use and the needed software will be pre-installed on a provided tablet.
* An electronic questionnaire will be used to induce subjects to follow the study procedures and to assess compliance afterwards.
* The heart rate and physical activity tracker will help determining if the subjects have followed the recommendation to avoid intense exercise in concomitance with the PPGR measurement
* A certain time flexibility is allowed to accommodate the participants' needs and reduce the risk of drop-outs.
* A conservative approach was used in the calculation of the sample size to reduce the risk of the study being underpowered in case of unexpected drop-out rate.
* The Metabolic Unit staff will be reachable, during working hours, by the participants to provide technical support and to monitor their safety.
* The study staff will be alerted via email every time that an adverse event is imputed in the adverse event collection tool.

The two products selected as positive and negative control for the present research project. Comparison of PPGR data generated in the present research project with existing data will allow evaluating the reliability of the remote approach compared to the traditional one.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participant
* Healthy status (based on anamnesis)
* Age between 18 and 45 years
* BMI between 18.5 and 29.9 kg/m2
* Able to understand and sign an informed consent form
* Able to respect the study procedures and timelines
* Swiss resident living in canton Fribourg (French part), Neuchâtel, Vaud and Valais which is in the competence of Ethical Committee of Vaud
* Having wireless internet access at home

Exclusion Criteria:

* Any known metabolic disease including diabetes or drug chronic intake (aspirin, vitamin C and mineral supplements, steroids, protease inhibitors, antidepressants, anxiolytic, or antipsychotics…) possibly impacting (to the opinion of the medical responsible): The digestion or absorption of nutrients, the postprandial glucose response
* Major medical/surgical event requiring hospitalization in the last 3 months
* Pregnancy or lactation
* Known food allergy and intolerance
* Medically known cutaneous hypersensitivity to adhesives, silicon watch-strap and plasters
* Alcohol intake higher than 2 servings per day. A serving is 0.4 dl of strong alcohols, 1 dl of red or white wine, or 3 dl of beer.
* Smokers
* Participant having a hierarchical link with the research team members

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-11-29 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-02-18 (Actual)

PRIMARY OUTCOMES:
Incremental area under the concentration curve (iAUC 0 to 120 minutes) of post-prandial glucose | From 0 (product intake) to 120 minutes
  Incremental area under the concentration curve (iAUC 0 to 120 minutes) of post-prandial glucose in the interstitial subcutaneous fluid as measured by a continuous glucose monitoring (Flash Glucose Monitoring FGM) commercial device (Abbott Freestyle Libre), as absolute values or as relative value to the raise observed for a glucose syrup as positive control and a resistant dextrin containing a non-digestible fiber as negative control

SECONDARY OUTCOMES:
Maximum concentration (Cmax) of post-prandial glucose | From 0 (product intake) to 120 minutes
  Maximum concentration (Cmax) of post-prandial glucose in the interstitial subcutaneous fluid as measured by FGM device
Time of Cmax (Tmax) of post-prandial glucose | From 0 (product intake) to 120 minutes
  Time of Cmax (Tmax) of post-prandial glucose in the interstitial subcutaneous fluid as measured by FGM device
Adverse events | Through subject participation, up to 2 weeks
  Incidence, type, severity and relation to the research product of possible adverse events experienced by the participants during the study
Gastro-intestinal tolerability | Through subject participation, up to 2 weeks
  Gastro-intestinal tolerability as assessed by visual analogue scale for the following symptoms: 1) Abdominal discomfort, 2) Decreased appetite, 3) Gastric reflux, 4) Nausea, 5) Diarrhea, 6) Headache
Heart rate | Through subject participation, up to 2 weeks
  Continuous heart rate measure (recorded by wearable activity tracker)
Physical activity | Through subject participation, up to 2 weeks
  Continuous physical activity measure (recorded by wearable activity tracker)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Sun, MD, Principal Investigator — Nestlé Research - Clinical Research Unit - Clinical Innovation Lab
Locations (1):
- Nestlé Research - Clinical Research Unit - Clinical Innovation Lab, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No